CLINICAL TRIAL: NCT00100542
Title: Psychiatric Co-Morbidity in Perinatally HIV-Infected Children and Adolescents
Brief Title: Psychiatric Problems in Children and Adolescents Infected With HIV at Birth
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Wende Levy, IMPAACT
Other Study IDs: PACTG P1055; U01AI068632 (NIH)
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: HIV Infections; Mental Disorders
Keywords: Treatment Experienced; Treatment Naive; Psychopathology; Anti-Retroviral Agents; Child; Adolescent
MeSH Terms: conditions — HIV Infections; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: All HIV infected and uninfected participants and their caregivers.
  Interventions: Behavioral: Psychiatric interviews

INTERVENTIONS:
Behavioral: Psychiatric interviews — Measures and questionnaires regarding mental health, pain, and adherence to treatment. No actual treatment or intervention is given as part of this study.

SUMMARY:
The purpose of this study is to determine whether HIV and anti-HIV drugs cause mental health problems or make mental health problems worse in children and adolescents who were infected with HIV at birth.

DETAILED DESCRIPTION:
Research has shown that HIV is able to penetrate the blood-brain barrier and may significantly affect the central nervous system (CNS). Although the effects of HIV on the CNS are not fully understood, there is growing evidence that the effects are psychosocial in nature; HIV infected children experience higher rates of psychiatric symptoms and hospitalizations than their uninfected counterparts. Confounding the HIV CNS relationship is evidence suggesting that the CNS effects of HIV may also be related to antiretroviral treatment. This study will examine the rates and severity of psychiatric symptoms in both HIV infected and uninfected children and adolescents. In addition, this study will determine the relationship between duration of antiretroviral treatment and psychiatric symptoms.

No treatment will be given as part of this study. The study will last for 96 weeks and be divided into two parts. In Part 1, HIV infected and uninfected participants and their caregivers will complete a series of measures and questionnaires regarding mental health, pain, and adherence to treatment. In Part 2, all participants and their caregivers will complete a subset of the original measures at Weeks 48 and 96. This follow-up part of the study will assess any long-term changes in psychiatric symptoms. In addition, a subset of HIV infected and uninfected participants and their caregivers will take part in psychiatric interviews at specified study sites. A portion of these interviews will be audio-taped.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Participants:

* Acquired HIV through mother-to-child transmission

Inclusion Criteria for HIV Uninfected Participants:

* HIV uninfected

Inclusion Criteria for All Participants:

* Living with same parent or primary caregiver for at least 12 months prior to study screening
* Willing and able to provide consent or assent

Exclusion Criteria for HIV Infected Participants:

* Acquired HIV through adult high-risk behavior, blood transfusion, or abuse

Exclusion Criteria for All Participants:

* IQ of 69 or lower, for participants whose primary language is English. More information on this criterion can be found in the protocol.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and their caregivers from specific clinics.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2005-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nachman, MD, Study Chair — Department of Pediatrics, Stony Brook University
Locations (32):
- United States (31):
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County Medical Center/USC, Los Angeles, California
  - UCLA Medical Center (Pediatric), Los Angeles, California
  - 4601 UCSD Mother, Child & Adolescent HIV Program, San Diego, California
  - UCSF, Moffitt Hospital (Pediatric), San Francisco, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Childrens Hospital (U. Colorado, Denver), Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Howard University Hospital, Washington D.C., District of Columbia
  - North Broward Hospital District, Fort Lauderdale, Florida
  - University of Florida - Health Science Center, Jacksonville, Florida
  - University of Miami (Pediatric), Miami, Florida
  - University of South Florida, St. Petersburg, Florida
  - Chicago Childrens Memorial Hospital (Pediatric), Chicago, Illinois
  - University of Maryland (Pediatric), Baltimore, Maryland
  - Childrens Hospital of Boston, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - New York University School of Medicine, New York, New York
  - Metropolitan Hospital Center, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - State University of New York at Stony Brook, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Duke University (Pediatric), Durham, North Carolina
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christophers Hosp. for Children, Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Memphis, Tennessee
  - Children's Hospital and Regional Medical Center/Seattle, Seattle, Washington
  - Northwest Family Ctr./Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Ctr., Seattle, Washington
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Background] Bachanas PJ, Kullgren KA, Schwartz KS, Lanier B, McDaniel JS, Smith J, Nesheim S. Predictors of psychological adjustment in school-age children infected with HIV. J Pediatr Psychol. 2001 Sep;26(6):343-52. doi: 10.1093/jpepsy/26.6.343. PMID 11490035
- [Background] De Luca A, Ciancio BC, Larussa D, Murri R, Cingolani A, Rizzo MG, Giancola ML, Ammassari A, Ortona L. Correlates of independent HIV-1 replication in the CNS and of its control by antiretrovirals. Neurology. 2002 Aug 13;59(3):342-7. doi: 10.1212/wnl.59.3.342. PMID 12177366
- [Background] Gaughan DM, Hughes MD, Oleske JM, Malee K, Gore CA, Nachman S; Pediatric AIDS Clinical Trials Group 219C Team. Psychiatric hospitalizations among children and youths with human immunodeficiency virus infection. Pediatrics. 2004 Jun;113(6):e544-51. doi: 10.1542/peds.113.6.e544. PMID 15173535
- [Background] Lwin R, Melvin D. Paediatric HIV infection. J Child Psychol Psychiatry. 2001 May;42(4):427-38. PMID 11383959
- [Background] Mellins CA, Smith R, O'Driscoll P, Magder LS, Brouwers P, Chase C, Blasini I, Hittleman J, Llorente A, Matzen E; NIH NIAID/NICHD/NIDA-Sponsored Women and Infant Transmission Study Group. High rates of behavioral problems in perinatally HIV-infected children are not linked to HIV disease. Pediatrics. 2003 Feb;111(2):384-93. doi: 10.1542/peds.111.2.384. PMID 12563068
- [Result] Chernoff M, Nachman S, Williams P, Brouwers P, Heston J, Hodge J, Di Poalo V, Deygoo NS, Gadow KD; IMPAACT P1055 Study Team. Mental health treatment patterns in perinatally HIV-infected youth and controls. Pediatrics. 2009 Aug;124(2):627-36. doi: 10.1542/peds.2008-2441. Epub 2009 Jul 13. PMID 19596734
- [Derived] Nachman S, Chernoff M, Williams P, Hodge J, Heston J, Gadow KD. Human immunodeficiency virus disease severity, psychiatric symptoms, and functional outcomes in perinatally infected youth. Arch Pediatr Adolesc Med. 2012 Jun 1;166(6):528-35. doi: 10.1001/archpediatrics.2011.1785. PMID 22312169